CLINICAL TRIAL: NCT01502761
Title: Intra-arterial Magnesium Therapy: A Novel Platorm for Neuroprotectant Delivery in Acute Stroke
Brief Title: Intra-arterial Magnesium Administration for Acute Stroke
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No safety issues. Low enrollment secondary to negative stroke studies 2013
Sponsor: University of Southern California (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, William Mack, Assistant Professor of Neurosurgery, University of Southern California
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-11-00339
Record Dates: First submitted 2011-12-22; First posted 2012-01-02 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-07

CONDITIONS: Acute Stroke
Keywords: stroke; Magnesium; endovascular
MeSH Terms: conditions — Stroke | interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Regional Intra-arterial Magnesium 0.75g (Experimental): Regional Intra-arterial magnesium only 0.75 mg Magnesium Sulfate (50% Total Dose): 5 patients
  Interventions: Drug: Magnesium Sulfate
- Regional Intra-arterial magnesium 1.5g (Experimental): Regional Intra-arterial magnesium Sulfate Only 1.5g (100% TD): 5 patients
  Interventions: Drug: Magnesium Sulfate
- Regional/ Distal (75/25%) Magnesium 1.5g (Experimental): Regional/ Distal intra-arterial magnesium (75% TD regional- 1.125g / 25% distal-0.375g): 5 patients
  Interventions: Drug: Magnesium Sulfate
- Regional/ Distal (50/50%) Magnesium 1.5g (Experimental): Regional/ Distal intra-arterial magnesium (50% TD regional- 0.75g/ 50% distal-0.75g): 5 patients
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — Intra-arterial

SUMMARY:
Stroke is the second leading cause of death and the leading cause of adult disability worldwide. This investigation will address the safety and feasibility of directed, intra-arterial Magnesium measurement and therapy, through endovascular access, in acute stroke patients. The proposal represents the first study to directly quantify levels of a systemically administered neuroprotectant in the region of cerebral ischemia. It also establishes a novel endovascular platform for direct delivery of neuroprotective agents to ischemic cerebral tissue distal to an occlusive thrombus. This research seeks to improve patient care by establishing a novel delivery mechanism for the rescue of threatened brain parenchyma that can be administered rapidly following acute stroke. If successful, this selective distribution will allow delivery to "at risk" tissue in a rapid manner. Salvage of viable, but threatened, penumbral tissue could afford stroke patients an increased probability of favorable long term outcome. The investigators hypothesize that endovascular, intra-arterial, Magnesium administration will deliver high concentration of this neuroprotective agent to otherwise inaccessible cerebral territories, while limiting systemic concentrations. The proposed investigation will evaluate the safety and feasibility of this novel treatment technique

ELIGIBILITY:
Inclusion Criteria:

1. Patient with acute cerebral ischemia due to ICA or MCA occlusion,
2. Patient's clinical attending physician plans mechanical embolectomy procedure as part of routine clinical care.
3. Age 21-95.

Exclusion Criteria:

1. Severe renal impairment with creatinine 3.0 or higher,
2. Myasthenia gravis,
3. Second or third degree heart block without a pacemaker in place,
4. Technical inability to navigate microcatheter to target clot,
5. Patient already enrolled in another experimental treatment trial. Exclusion criteria 1-3 are all contraindications to magnesium therapy.

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J Mack, MD, Principal Investigator — University of Southern California; Jeffrey Saver, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - University California Los Angeles: Ronald Reagan and Santa Monica Hospitals, Los Angeles, California
  - University of Southern California University and LA County Hospitals, Los Angeles, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Regional Intra-arterial Magnesium 0.75g: Regional only 0.75 mg Magnesium Sulfate (50% Total Dose): 5 patients
  Magnesium Sulfate: Intra-arterial
- Regional/ Distal (75/25%) Magnesium 1.5g: Regional/ Distal(75% TD regional- 1.125g / 25% distal-0.375g): 5 patients
  Magnesium Sulfate: Intra-arterial
- Regional/ Distal (50/50%) Magnesium 1.5g: Regional/ Distal (50% TD regional- 0.75g/ 50% distal-0.75g): 5 patients
  Magnesium Sulfate: Intra-arterial
Period: Overall Study
Arm/Group | Regional Intra-arterial Magnesium 0.75g | Regional Intra-arterial Magnesium 1.5g | Regional/ Distal (75/25%) Magnesium 1.5g | Regional/ Distal (50/50%) Magnesium 1.5g
Started | 4 | 0 | 0 | 0
Completed | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 4 patients were enrolled (regional intra-arterial Magnesium 0.75g) before the study was stopped (not due to safety concerns). They were all enrolled in the first group
Groups:
- Total: Total of all reporting groups
Arm/Group | Regional Intra-arterial Magnesium 0.75g | Regional Intra-arterial Magnesium 1.5g | Regional/ Distal (75/25%) Magnesium 1.5g | Regional/ Distal (50/50%) Magnesium 1.5g | Total
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.25 (13.25) |  |  |  | 68.25 (13.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  |  |  | 2
  Male | 2 |  |  |  | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  |  | 0
  Asian | 0 |  |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  |  | 0
  Black or African American | 0 |  |  |  | 0
  White | 4 |  |  |  | 4
  More than one race | 0 |  |  |  | 0
  Unknown or Not Reported | 0 |  |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 |  |  |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Magnesium Concentration in Region of Cerebral Ischemia
Description: Peripheral Magnesium Levels, meq/L will be obtained through the femoral sheath at the beginning (baseline) and end (post-treatment) of each case. These will be averaged to obtain a femoral Magnesium level. Magnesium levels distal to the occlusion will be measured at the first pass of the clot retrieving device.
Time Frame: Mg level: 1) Peripheral: Baseline and post-treatment (averaged); 2) Distal: after first pass of the clot retriever
Population: Enrollment only occurred in the first arm (lowest dose) of the study as the arms were planned to enroll sequentially. The study was not stopped due to safety concerns
Measure: Mean (Standard Deviation); unit: meq/L
Arm/Group | Regional Intra-arterial Magnesium 0.75g | Regional Intra-arterial Magnesium 1.5g | Regional/ Distal (75/25%) Magnesium 1.5g | Regional/ Distal (50/50%) Magnesium 1.5g
Number analyzed (Participants) | 4 | 0 | 0 | 0
meq/L
  Distal Mg level | 1.475 (.3403) |  |  |
  Peripheral Mg level | 1.513 (.2462) |  |  |

2. Secondary Outcome: Number of Participants With Procedure Related Serious Adverse Event
Description: Periprocedural clinical, radiographic and laboratory data will be collected and analyzed to detect Mg related adverse events. Outcome will be assessed perioperatively and at 24 hours, 30 days (+/- 10 days) and 90 days (+/- 15 days)
Time Frame: intraprocedure, postoperative day 1, 1 month, 3 month
Measure: Count of Participants; unit: Participants
Arm/Group | Regional Intra-arterial Magnesium 0.75g | Regional Intra-arterial Magnesium 1.5g | Regional/ Distal (75/25%) Magnesium 1.5g | Regional/ Distal (50/50%) Magnesium 1.5g
Number analyzed (Participants) | 4 | 0 | 0 | 0
Participants | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Regional Intra-arterial Magnesium 0.75g | Regional Intra-arterial Magnesium 1.5g | Regional/ Distal (75/25%) Magnesium 1.5g | Regional/ Distal (50/50%) Magnesium 1.5g
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 2/4 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regional Intra-arterial Magnesium 0.75g (N=4) | Regional Intra-arterial Magnesium 1.5g (N=0) | Regional/ Distal (75/25%) Magnesium 1.5g (N=0) | Regional/ Distal (50/50%) Magnesium 1.5g (N=0)
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parotiditis with sepsis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regional Intra-arterial Magnesium 0.75g (N=4) | Regional Intra-arterial Magnesium 1.5g (N=0) | Regional/ Distal (75/25%) Magnesium 1.5g (N=0) | Regional/ Distal (50/50%) Magnesium 1.5g (N=0)
Cerebral Edema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischemic change on brain imaging (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhagic Transformation of stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sick Sinus Syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
increased blood glucose (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was terminated early (with enrollment only in the first arm) by the investigators due to low enrollment (given results of relevant studies at the time) . There were no safety concerns with the trial or the agent.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No